CLINICAL TRIAL: NCT02202291
Title: Prospective Multicenter Study on the Identification of Genetic Abnormalities Predisposing to Vasospasm From a Privileged Model: the Primary Raynaud's Phenomenon
Acronym: RAY-GENE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: RC14_0086; 2014-A00470-47 (Other: ANSM)
Record Dates: First submitted 2014-07-15; First posted 2014-07-29 (Estimated); Last update posted 2020-06-24 (Actual); Status verified 2020-06

CONDITIONS: Primary Raynaud's Phenomenon (PR); Genetic Mutations Causing PR; Study of Patients and Their Relatives (With or Without Primary PR)
Keywords: Raynaud's phenomenon, Vasospasm, Genetics
MeSH Terms: conditions — Raynaud Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Patient with Raynaud's phenomenon (Experimental)
  Interventions: Genetic: Demonstration of genetic mutations causing Raynaud's phenomenon

INTERVENTIONS:
Genetic: Demonstration of genetic mutations causing Raynaud's phenomenon — Such an approach allows to highlight chromosomal regions shared only by individuals within a family and thus highlight the genetic mutations causing the Raynaud phenomenon . The ultimate goal is to identify new pathways involved in vasospasm.
  Patients with primary Raynaud phenomenon will be identified during a consultation of vascular medicine and internal medicine in one of the centers participating to the study. Those patients with a primary PR will be considered as Index cases.
  The investigators will conduct genealogical trees of index cases to identify families, whose number of healthy individuals and those with relevant PR makes sense for a family genetic study, i.e. a genetically informative family.
  Other Names: Recruitment of familial forms of Raynaud phenomenon (patients with primary; Raynaud phenomenon and their relatives) to perform genetic analysis of; exome sequencing type combined with an analysis of family bonding.

SUMMARY:
Vasospasm is a transient contraction causing a decrease in caliber of a vessel and thus a decrease in vascularization in a vascular territory leading to suffering of tissue in the sector concerned. Vasospasm-related diseases have different clinical presentations such as migraine, spastic angina, hypertension related to vasospasm or primary Raynaud's phenomenon (RP). These diseases have few therapeutic methods due to poorly understood pathophysiology. For migraine and angina, the vascular exploration is problematic unlike for primary Raynaud's phenomenon (RP).

Primary Raynaud's phenomenon (RP) is a common peripheral vascular disease to cold with an estimated prevalence between 5-9 % of the general population. It is the expression of an extreme vasospasm microcirculation of the extremities linked to hypersensitivity to cold and that is clinically expressed by the occurrence of syncope stages where the fingers are anesthetized and white, followed by a stage with hyperemic restaining .

The objective of our study is to identify new metabolic pathways involved in vasospasm in order to consider new specific treatments, currently lacking.

The identification of these pathways will be made by the detection of genetic abnormalities causing vasospasm in Raynaud's phenomenon. This disease is a perfectly appropriate model to study vasospasm by its high frequency in the population, its hereditary nature and simple diagnosis. The powerful current genetic strategies will be applied to this model (exome sequencing combined to family connection analysis).

DETAILED DESCRIPTION:
Patients with primary Raynaud phenomenon will be identified during a consultation of vascular medicine and internal medicine in one of the centers participating to the study. Those patients with a primary PR will be considered as Index cases.

In all participating centers, there will be a recruitment of index cases without family screening to form a series of cases that will validate the results obtained in family forms.

The investigators will conduct genealogical trees of index cases to identify families, whose number of healthy individuals and those with relevant PR makes sense for a family genetic study, i.e. a genetically informative family.

In all centers, relatives of included Index cases, agreeing to participate in this research, will be enrolled and followed.

Nantes University Hospital is the only center to perform a cold test (for reasons of availability of the technique) but this test will be reserved for patients whose diagnosis of primary Raynaud's phenomenon would be doubtful. Exposed identified relatives, agreeing to participate in this research, will all be included and followed in their enrollment center.

ELIGIBILITY:
Inclusion criteria:

* Major Subject (age ≥ 18 years)
* Index case with all the diagnostic criteria for primary Raynaud phenomenon, according to current recommendations OR Related index case (relatives' patients) with or without a primary Raynaud phenomenon.
* Written consent to participate in the study
* Written consent to participate in the collection of biological samples

Exclusion criteria:

* Subjects who have expressed their inability or refusal to sign an informed consent,
* Index case with a secondary Raynaud phenomenon (suspected by clinical examination and confirmed by capillaroscopy and laboratory tests: antinuclear antibody, abnormalities of capillaroscopy mégacapillaire dystrophy or other major deviation).

(Criterion not applicable to related parties, i.e. family members of Index cases)

- Pregnant Woman.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 258 (Actual)
Dates: Start 2014-10-13 (Actual); Primary Completion 2020-06-10 (Actual); Study Completion 2020-06-10 (Actual)

PRIMARY OUTCOMES:
To identify number of genes involved in vasospasm of primary Raynaud's phenomenon (RP) and determine the genetic cause of primary RP | 36 months
  Patients with primary Raynaud's phenomenon and their relatives will be recruited to establish familial forms of Raynaud's phenomenon. This will allow perform genetic analysis using new approaches to genetic broadband (exome sequencing analysis + linkage analysis). This approach will allow specify which chromosomal regions are shared only by affected individuals, and identify new candidate genes

SECONDARY OUTCOMES:
To determine number of phenotypes associated to genotype of primary Raynaud's phenomenon | 36 months
  Based on the identified genes in different families, a descriptive analysis will allow associate them with different RP phenotypes (isolated RP or RP associated with migraines, angina or hypertension) and risk factors.

CONTACTS AND LOCATIONS:
Overall Officials: Marc-Antoine Pistorius, Prof, Study Director — University Hospital of Nantes; Marc-Antoine Pistorius, Prof, Principal Investigator — University Hospital of Nantes; Luc Bressollette, Prof, Principal Investigator — University Hospital of Brest; Patrick Jégo, Prof, Principal Investigator — University Hospital of Rennes; Samir Henni, Dr, Principal Investigator — University Hospital of Angers; Jean-Manuel Kubina, Dr, Principal Investigator — Hospital of La Roche/Yon; Pierre Plissonneau Duquene, Dr, Principal Investigator — Hospital of St Nazaire
Locations (6):
- France (6):
  - CHU Angers - Service d'Explorations vasculaires, Angers
  - CHRU HOPITAL CAVALE BLANCHE - Service de Médecine vasculaire, Brest
  - CHD La Roche sur Yon - Service Angéiologie, La Roche-sur-Yon
  - CHU de NANTES - Service de Médecine Interne, Nantes
  - C.H.R. HOPITAL SUD - Service de Médecine interne, Rennes
  - Ch Saint Nazaire, Saint-Nazaire

IPD SHARING:
Plan to Share IPD: No